CLINICAL TRIAL: NCT03871114
Title: Evaluation of Salivary Levels of miR-155 and IL-10 in Oral Lichen Planus Patients Before and After Treatment With Topical Corticosteroid
Brief Title: Evaluation of Salivary Level of miR-155 and IL-10 in Oral Lichen Planus Patients Before and After Treatment With Topical Corticosteroid
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Amr, Associate Professor, Cairo University
Other Study IDs: miR-155 OLP
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide; Orabase; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OLP patients: fifteen patients with atrophic /erosive OLP will receive treatment with topical triamcinolone acetonide in orabase 1mg/g 3 times /day and assessed every week for 4 weeks
  Interventions: Drug: Triamcinolone Acetonide in orabase
- Control group

INTERVENTIONS:
Drug: Triamcinolone Acetonide in orabase — treatment of OLP with topical steroid
  Other Names: topical corticosteroid
  Groups: OLP patients

SUMMARY:
Thirty patients will be recruited from the outpatient clinic of the faculty of dentistry.fifteen systemically healthy individuals with normal mucosa and fifteen atrophic/erosive oral lichen planus patients. Oral lichen planus patients will be treated with a topical steroid and miR-155 and IL-10 will be assessed in saliva before and after 4 weeks of topical steroids use

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically and histopathologically diagnosed as having atrophic/erosive OLP.
* Patients free from any other oral lesions
* cooperative patients who agrees to take the supplied medications.
* Patients who are systemically healthy

Exclusion Criteria:

* Patients suffering from any systemic disease.
* Treatment with any systemic treatment such as systemic steroids, other immunosuppressive drugs or non-steroidal anti-inflammatory drugs at least eight weeks.
* Treatment with any oral topical medications for at least four weeks prior to the study.
* Pregnant and lactating women.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with atrophic/erosive oral lichen planus
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Measurement of salivary levels of miR-155 in OLP before treatment | baseline
  assessment of miR-155 in saliva of patients with OLP before treatment
Measurement of salivary levels of IL-10 in OLP before treatment | baseline
  assessment of IL-10 in saliva of patients with OLP before treatment

SECONDARY OUTCOMES:
Measurement of salivary levels of miR-155 in OLP after treatment | 4 weeks
  assessment of miR-155 in saliva of patients with OLP after treatment
Measurement of salivary levels of IL-10 in OLP after treatment | 4 weeks
  assessment of IL-10 in saliva of patients with OLP after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt